CLINICAL TRIAL: NCT04091932
Title: The Effect and Safety of Programmed Cell Death Protein 1 (PD-1) Inhibitor on AIDS Patients With Progressive Multifocal Leukoencephalopathy (PML): A One-center, Single-arm and Prospective Study
Brief Title: Treatment of PD-1 Inhibitor in AIDS-associated PML
Acronym: TPAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-57
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Progressive Multifocal Leukoencephalopathy; AIDS
Keywords: PD-1 inhibitor; Pembrolizumab; Progressive Multifocal Leukoencephalopathy; AIDS
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal; Acquired Immunodeficiency Syndrome | interventions — pembrolizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab treatment (Experimental): Pembrolizumab dosage form:100mg/4ml dosage:2mg/kg weight frequency: once per 4 weeks duration:12 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Monthly usage of Pembrolizumab (2mg/kg weight) for 3 months.
  Other Names: PD-1 inhibitor

SUMMARY:
PD-1 inhibitor （Pembrolizumab, 2mg/kg weight, once per 4 weeks and 3 times of medication usage）treatment on AIDS patients with progressive multifocal leukoencephalopathy.

DETAILED DESCRIPTION:
This is a one-center, single-arm and prospective study, planing recruiting 10 AIDS-associated PML patients. All patients will receive PD-1 inhibitor (Pembrolizumab) for 12 weeks, and the dose for each time is 2 mg per kg/weight, and the frequency is once per 4 weeks. The effect and safety of Pembrolizumab on AIDS-associated PML will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65
2. Diagnosed of HIV by lab confirmation
3. Diagnosed of PML by diplomatic radiologists through brain MRI or by brain biopsy once there are some concerns on radiologic diagnosis.
4. agree to sign the consent
5. agree to use contraception measures during 4 weeks before to 6 months after this study

Exclusion Criteria:

1. Pregnancy or lactating women or planing birth during this study
2. Anticipated bad treatment compliance
3. Within 6 months before joining this study, receive other immunosuppressors, immunomodulators or cytotoxic drugs (glucocorticoid is allowed)；
4. With neutrophil<1000/mm3 or platelet<75000/mm3 or allergic to PD-1 inhibitor 5）With severe basic diseases in heart, brain, lung, liver, kidney

6) disagree to sign the consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the rate of non-progressors and recovers of AIDS patients with PML in 6 months after receiving PD-1 inhibitor | 6 months
  With treatment of Pembrolizumab for 6 months, we will evaluate the rate of non-progressors and recovers of AIDS patients with PML
the rate of non-progressors and recovers of AIDS patients with PML in 12 months after receiving PD-1 inhibitor | 12 months
  With treatment of Pembrolizumab for 12 months, we will evaluate the rate of non-progressors and recovers of AIDS patients with PML

SECONDARY OUTCOMES:
the negative conversion rate of John Cunningham virus (JCV) in cerebrospinal fluid，blood and urine in patients receiving Pembrolizumab. | 3 months
  With treatment of Pembrolizumab for 3 months, we will evaluate the negative conversion rate of JCV in cerebrospinal fluid，blood and urine
Side effects associated with Pembrolizumab | 12 months
  To investigate the safety of Pembrolizumab in HIV patients
The rate of patients with decreased HIV viral reservoir | 12 months
  To investigate the rate of patients with decreased HIV viral reservoir

CONTACTS AND LOCATIONS:
Overall Officials: Biao Zhu, PhD, Principal Investigator — Zhejiang University
Locations (1):
- the first affiliated hospital of Zhejiang university school of medicine, Hangzhou, Zhejiang, China